CLINICAL TRIAL: NCT05561920
Title: Dependencies of Acoustic Signal and Image Recordings of Phonatory Movement of the Pharyngoesophageal Mucosa in Laryngectomy Patients Using High-speed Video Endoscopy and a Biomechanical Model
Brief Title: Phonatory Movement of the Pharyngoesophageal Mucosa in Laryngectomy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-HS camera
Record Dates: First submitted 2022-09-15; First posted 2022-09-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Larynx Cancer; Laryngectomy; Status
Keywords: Laryngectomy; Endoscopy; Speech,acoustics; High speed imaging; Speech,alaryngeal; Pharyngoesophageal segment; Biomechanics model
MeSH Terms: conditions — Laryngeal Neoplasms; Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult laryngectomised patients: Patients who have undergone total laryngectomy and completed minimal their 6-month period without disease after surgery and post-operative treatments such as radiotherapy or chemotherapy
  Interventions: Device: High - speed video endoscopy (HSV); Device: Acoustic voice analysis; Behavioral: Quality of life questionnaire

INTERVENTIONS:
Device: High - speed video endoscopy (HSV) — Describe anatomical and morphological characteristics o phonatory movement of PEM in laryngectomy patients
Device: Acoustic voice analysis — acoustic program (lingWAVES - Voice and speech analyser) - measuring the values of acoustic parameters in voice recordings
Behavioral: Quality of life questionnaire — Filling out questionnaires

SUMMARY:
Therapy of advanced cancer of the larynx includes excision of the entire larynx. After the removal of the larynx, the pharyngoesophageal segment (PES) is created by reconstruction of the soft tissue of the pharynx and oesophagus, and its vibration creates a replacement voice. High-speed video endoscopy (HSV) is the only method that visualizes and measures vibration of pharyngoesophageal mucosa (PEM) after laryngectomy. Acoustic characteristics of three forms of the rehabilitated voice of laryngectomized persons (oesophageal voice, tracheoesophageal voice using a speech prosthesis and electrolarynx) have been satisfactorily described but, the interdependence of acoustic and visual representations of the phonatory movement of the PES is still insufficiently investigated. In recent years, the development of biomechanical models is created to analyse the vibration of the PES, but still no uniform results have been achieved that would explain whether the parameters obtained from the analysis of the waveform of the PES can be compared with the parameters obtained from the acoustic analysis of the voice of a laryngectomized patients

DETAILED DESCRIPTION:
The first aim of this study is to describe phonatory movement of PEM in laryngectomy patients with HSV and then with biomechanical model, analyse these recordings and examine relationship between the obtained parameters and the parameters obtained using the acoustic analysis of the voice of a laryngectomized person. Secondary aim is to assess the impact of loss of voice in terms of psychological and socioeconomic problems in laryngectomy patients using Croatian version of the Self-Evaluation of Communication Experiences after Laryngectomy (SECEL:HR) questionnaire and to examine whether there is a connection between the parameters obtained from the analysis of acoustic recordings and HSV recordings with the results of the questionnaire i.e., with better or worse postoperative adaptation and satisfaction with the replacement voice.

This is a non-interventional, prospective study of laryngectomised participants who completed oncological treatment and underwent voice rehabilitation. The data will be collected at the Clinical Department for Otorhinolaryngology and Head and Neck Surgery - University Hospital Centre, Osijek, Clinical Department for Otorhinolaryngology and Head and Neck Surgery - University Hospital Centre, Zagreb.

In the first phase of the research, translation and cultural adaptation of a Croatian version of the SECEL questionnaire will be carried out ( ClinicalTrials.gov Identifier: NCT05346237).

Second phase will enrol approximately 50 laryngectomised participants independent from the first phase of research. Data on surgical and oncological treatment, voice rehabilitation method, comorbidities and drug therapy will be collected retrospectively from the patient's medical histories. Ear,nose and throat examination and endoscopic evaluation of swallowing will be performed in order to rule out the presence of non-eligibility criteria. All subjects will fill out a validated questionnaire in Croatian (SECEL:HR). Voice production time will be measured, and subjects will undergo acoustical voice assessment and HSV during voice production. The visualisation of the pharyngoesophageal segment itself will be analysed - phase closure, pharyngoesophageal segment shape (circular, triangular, split side to side, split anterior-posterior, irregular), then the presence and location of visible vibration, and the presence of a mucosal wave. For the processing of HSV videos a computer program will be developed. Based on the collected data, the parameters of the assumed multi-mass coupled biomechanical model will be identified and compared with the acoustic recording of each respondent.

ELIGIBILITY:
Inclusion Criteria:

* laryngectomised patients who completed minimal their 6-month period without disease after surgery and post-operative treatments such as radiotherapy or chemotherapy
* patients with preserved reading skills
* regular presence at follow-up visits

Exclusion Criteria:

* age less than 18 years
* acute respiratory infection of the upper or lower respiratory tract
* other primary cancer in the upper aerodigestive tract or lung
* presence of neurologic or pulmonary diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult male laryngectomised patients who completed oncological treatment and underwent voice rehabilitation
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
High speed video endoscopy recordings | 15 minutes for each participants
  Visual recording of the mucosa of the pharyngoesophageal segment will be performed with High speed video endoscopy (Wolf 5562 ENDOCAM) during the phonation of the letter "a". Recording is performed through the mouth with a rigid endoscope connected to an High speed camera.
Acoustic analysis | 15 minutes
  acoustic program- measuring the quality of voice each laryngectomised patients during phonation of vowel "a". Voice recordings will be analysed in the acoustic program (lingWAVES - Voice and speech analyser)
Maximum phonation time | 2 minutes
  Measurement of the longest possible relaxed phonation of the voice "a" by a speech therapist
Croatian version of the SECEL (SECEL:HR) questionnaire. | 15 minutes
  Completing the Croatian version of the SECEL questionnaire. Questionnaire consists of two parts. The first part examines the relevant general data on the person filling out the questionnaire, while the second part consists of 35 items questionably or statement-designed to examine communication experiences. Patients estimates the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always)
Development of Biomechanical model for vibration analysis obtained by High - speed video endoscopy | 3 months
  The development of the biomechanical model of the PES in order to quantify non-stationary PE-vibrations and drawing conclusions on the temporal characteristics of tissue stiffness, oscillating mass, pressure, and geometric distributions within the PE-segment. Biomechanical model will identify mathematical dependencies and analyse extracted time signals of the PES opening and contours which will compare video spectral analysis from high- speed video endoscopy imaging and the parameters obtained using the acoustic analysis of the voice of a laryngectomized person.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Đanić Hadžibegović, Assoc. Prof, Study Chair — Clinical Hospital Centre Zagreb; Andrijana Včeva, Full Prof, Study Chair — University Hospital Osijek
Locations (1):
- University Hospital Osijek, Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zenga J, Goldsmith T, Bunting G, Deschler DG. State of the art: Rehabilitation of speech and swallowing after total laryngectomy. Oral Oncol. 2018 Nov;86:38-47. doi: 10.1016/j.oraloncology.2018.08.023. Epub 2018 Sep 12. PMID 30409318
- [Background] van As CJ, Tigges M, Wittenberg T, Op de Coul BM, Eysholdt U, Hilgers FJ. High-speed digital imaging of neoglottic vibration after total laryngectomy. Arch Otolaryngol Head Neck Surg. 1999 Aug;125(8):891-7. doi: 10.1001/archotol.125.8.891. PMID 10448737
- [Background] Schwarz R, Huttner B, Dollinger M, Luegmair G, Eysholdt U, Schuster M, Lohscheller J, Gurlek E. Substitute voice production: quantification of PE segment vibrations using a biomechanical model. IEEE Trans Biomed Eng. 2011 Oct;58(10):2767-76. doi: 10.1109/TBME.2011.2151860. Epub 2011 May 10. PMID 21558056
- [Background] Huttner B, Luegmair G, Patel RR, Ziethe A, Eysholdt U, Bohr C, Sebova I, Semmler M, Dollinger M. Development of a time-dependent numerical model for the assessment of non-stationary pharyngoesophageal tissue vibrations after total laryngectomy. Biomech Model Mechanobiol. 2015 Jan;14(1):169-84. doi: 10.1007/s10237-014-0597-1. Epub 2014 May 27. PMID 24861998
- [Background] Schlegel P, Stingl M, Kunduk M, Kniesburges S, Bohr C, Dollinger M. Dependencies and Ill-designed Parameters Within High-speed Videoendoscopy and Acoustic Signal Analysis. J Voice. 2019 Sep;33(5):811.e1-811.e12. doi: 10.1016/j.jvoice.2018.04.011. Epub 2018 May 31. PMID 29861291
- [Background] Schindler A, Mozzanica F, Brignoli F, Maruzzi P, Evitts P, Ottaviani F. Reliability and validity of the Italian self-evaluation of communication experiences after laryngeal cancer questionnaire. Head Neck. 2013 Nov;35(11):1606-15. doi: 10.1002/hed.23198. Epub 2012 Nov 20. PMID 23169480
- [Background] Debruyne F, Delaere P, Wouters J, Uwents P. Acoustic analysis of tracheo-oesophageal versus oesophageal speech. J Laryngol Otol. 1994 Apr;108(4):325-8. doi: 10.1017/s0022215100126660. PMID 8182320
- [Background] Dooks P, McQuestion M, Goldstein D, Molassiotis A. Experiences of patients with laryngectomies as they reintegrate into their community. Support Care Cancer. 2012 Mar;20(3):489-98. doi: 10.1007/s00520-011-1101-4. Epub 2011 Feb 6. PMID 21298450